CLINICAL TRIAL: NCT01709058
Title: Prospective, Randomized, Single Blind Trial on the Effects of Paravertebral Intramuscular Oxygen-ozone Therapy on Back Pain in Subjects Aged 65 or Older
Brief Title: Study on the Effects of Oxygen-ozone Therapy on Back Pain in Subjects Aged 65 or Older
Acronym: O2-O3
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Regione Marche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INRCA-02-2011; 2011-003185-33 (EudraCT Number)
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Back Pain
Keywords: Back Pain; Therapeutics; Aged; Injections, Intramuscular; Oxygen; Ozone; Geriatric Assessment; Trace Elements; Oxidative stress
MeSH Terms: conditions — Back Pain | interventions — Injections, Intramuscular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramuscular/paravertebral injections of Oxygen-Ozone (Experimental): This group will be treated with "Intramuscular/paravertebral injections of Oxygen-Ozone" twice a week for six weeks
  Interventions: Drug: Intramuscular/paravertebral injections of Oxygen-Ozone
- Simulated treatment (Other): The "Simulated intramuscular/paravertebral injections" will mimic the Oxygen-Ozone injections in the area to be treated by pricking the skin with the needle without drilling. These simulated injections will be performed twice a week for six weeks.
  Interventions: Other: Simulated intramuscular/paravertebral injections

INTERVENTIONS:
Drug: Intramuscular/paravertebral injections of Oxygen-Ozone — Medical Oxygen will be used as a part of the injected mixture (100% oxygen, 200 bar compressed gas in steel cylinder with valve 14 with an integrated reductive). For the generation of the Oxygen-Ozone mixture a certified equipment OZONOSAN alpha plus will be used according to the D.L. 46/97, EEC Directive 93/42, class 2A with a photometer. The mixture of O2-O3 is produced through a method called "silent discharge". Intramuscular/paravertebral injections to 3 cm from the spinal medial line will be performed introducing 5-20 mL of oxygen-ozone to each point, at a concentration of 10-20 micrograms/mL, for a total volume of 40 mL
  Other Names: oxygen-ozone treatment
  Arms: Intramuscular/paravertebral injections of Oxygen-Ozone
Other: Simulated intramuscular/paravertebral injections — The simulated treatment administration will mimic the treatment in the area to be treated by pricking the skin with the needle without drilling. A light massage will be practice by hand and the application area will be covered with a bandage adhesive leaving the patient in the prone position for 10-15 minutes.
  Arms: Simulated treatment

SUMMARY:
This study aims to evaluate the efficacy of the oxygen-ozone therapy in the treatment of back pain in subjects aged 65 or older. In particular, the intramuscular injection technique/paravertebral of oxygen-ozone mixture, a minimal invasive treatment with respect to intradiscal infiltration/intraforaminal technique, will be used.

DETAILED DESCRIPTION:
Back pain is a leading cause of disability, including impairment in activities of daily living. In particular, the persistence of low back pain is more frequent in the elderly, associated with functional limitations and difficulties to perform tasks in everyday life. In addition to pharmacological treatments, various non-surgical interventional procedures are used for the treatment of low back pain. Some recent studies have evaluated the interventional oxygen-ozone (O2-O3) therapy in the treatment of back pain. However, these results are based on the technique of intradiscal infiltration / intraforaminal of O2-O3, while the intramuscular injection technique / paravertebral is the most widely used in clinical practice in Italy. In general, minimally invasive treatments such as percutaneous infiltration, are well tolerated and have been shown to produce clinical results, although the number of controlled studies is still scarce and the studies are often not comparable. Taking into account the above considerations, it seems appropriate to try to broaden the knowledge on the use of O2-O3 in the treatment of low back pain, using the technique of intramuscular injection / paravertebral, with particular reference to the elderly population.

The primary objective of this trial is therefore to evaluate the effects of O2-O3 therapy in the treatment of back pain associated with lumbar disc disease using the technique of intramuscular injection/paravertebral. These effects will be evaluated after a 6 weeks treatment period and after a 3 months follow-up period.

The project will include 130 subjects aged 65 or older who will be randomly enrolled in two different types of intervention:

* Oxygen-ozone therapy
* Simulated treatment

fully described below in the section: Interventions

In addition to clinical evaluations, the trial will contribute to the study of biological bases of the O2-O3 therapy as the levels of trace elements, oxidative status and antioxidant capacity in plasma will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 or older
* intervertebral disc degeneration
* back pain persistent for at least 6 weeks
* painkillers and anti-inflammatory drugs
* ODI score at baseline between 30 and 80%

Exclusion Criteria:

* heart failure
* favism
* clinically hyperthyroidism
* cancer and concomitant chemo-or radio-therapy
* epilepsy
* asthma
* life expectancy of 6 months or less
* psychotic drugs
* clinical signs of radiculopathy
* polyradiculopathy
* progressive neurological deficit
* lumbar stenosis
* spondylolisthesis
* diabetic neuropathy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index(ODI) | 6 weeks
  The Oswestry Disability Index (ODI) is used to investigate the functional impairment in activities of daily living related to low back pain. The ODI is one of the main measuring instruments necessary for the evaluation of disability from pain and is considered the gold standard for evaluation of disability in low back pain. It consists of 10 questions with multiple answers in which the patient chooses the answer that comes closest to its current state or to that of the last 2 weeks.
  Response to treatment is considered as a binary classification: "success" if the Oswestry Disability Index is between 0 and 20% (minimal disability) and "failure" in the other cases.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 3 months follow-up
  The Oswestry Disability Index (ODI) is used to investigate the functional impairment in activities of daily living related to low back pain. The ODI is one of the main measuring instruments necessary for the evaluation of disability from pain and is considered the gold standard for evaluation of disability in low back pain. It consists of 10 questions with multiple answers in which the patient chooses the answer that comes closest to its current state or to that of the last 2 weeks.
  Response to treatment is considered as a binary classification: "success" if the Oswestry Disability Index is between 0 and 20% (minimal disability) and "failure" in the other cases.
Comprehensive geriatric assessment by INTERRAI-MDS-HC/VAOR-ADI instrument | 6 weeks
  identification information, personal data at admission, assessment date, cognitive function, communication and vision, mood and behaviour, physical function, incontinence, diagnosis of the disease, health conditions, oral and nutrition status, skin conditions, medications, treatment and procedures, advanced directives, discharge potential, discharge, assessment information, anamnestic-clinical data, standardised clinical assessment, physical performance tests
intake of paracetamol | 6 weeks
  The use of paracetamol is allowed during the study period for the treatment of low back pain, at a dose of no more than 4 grams a day
oxidative stress | 6 weeks
  The evaluation of oxidative stress by the d-ROMs test and total antioxidant capacity by the anti-ROMs test will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- INRCA Hospital, via della Montagnola, 81, Ancona, Italy